CLINICAL TRIAL: NCT02282930
Title: An Open-Label Pilot Study of ACTH in the Treatment of IgA Nephropathy at High Risk of Progression
Brief Title: Pilot Study of ACTH in the Treatment of Immunoglobulin A (IgA) Nephropathy at High Risk of Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Fernando Fervenza, MD, PhD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-006965
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Progressive IgA Nephropathy; Proteinuria
Keywords: ACTH; Acthar; IgA; Progressive; Nephropathy; renal function
MeSH Terms: conditions — Proteinuria; Kidney Diseases | interventions — Adrenocorticotropic Hormone; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACTH Gel (Experimental): Injected does of 80 units subcutaneously twice weekly for 6 months.
  Interventions: Drug: ACTH (Acthar) Gel

INTERVENTIONS:
Drug: ACTH (Acthar) Gel — Injected dose of 80 units subcutaneously twice weekly for 6 months.

SUMMARY:
This study is designed to answer whether patients with progressive IgA nephropathy, who receive Acthar (ACTH) gel injection at a dose of 80 units subcutaneously twice weekly for 6 months is effective in inducing improvement in proteinuria and renal function.

ELIGIBILITY:
Inclusion:

* Proteinuria > 1000 mg/24h despite documented ACEi/ARB therapy and adequate blood pressure control for > 3 months.
* Quantified 24h creatinine clearance > 30 ml/min/1.73m2.
* Blood pressure < 130/80 mmHg at > 75% of the readings.
* Henoch Schoenlein Purpura (HSP): Patients with biopsy proven IgA nephropathy and clinical features consistent with Henoch Schonlein Purpura will be considered eligible for the study.
* Patient must be able to receive injections to be enrolled in the study.
* Patient must have a kidney biopsy slide on file - that can be sent to Mayo Clinic.

Exclusion:

* Clinical and histologic evidence of IgA predominant Lupus nephritis
* Patients with greater than 50% glomerular senescence or cortical scarring on renal biopsy.
* Serum Cr > 3.0 mg/dL or creatinine clearance glomerular filtration rate (GFR) < 30 ml/min at the time of screening
* Patients with history of Crohn's disease or Celiac Sprue
* Clinical evidence of cirrhosis, chronic active liver disease.
* Known infection with hepatitis B, hepatitis C, or HIV (Patients will be serologically screened prior to study entry (if the rest has been completed in the last two years, the patient will not have to undergo additional testing).
* Active systemic infection with bacterial, viral, fungal, or mycobacterial or atypical mycobacterial infections (excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Positive pregnancy test or breast feeding at time of study entry (urine pregnancy test will be performed for all women of childbearing potential no later than 7 days prior to treatment) or patients unwilling to comply with contraceptive measures as outlined above.
* Patients receiving therapy with oral prednisone or glucocorticoid equivalent in the past 3 months.
* Patients who had received immunosuppressive therapy including cyclophosphamide, mycophenolate mofetil (MMF), cyclosporine, tacrolimus or azathioprine in the last 6 months.
* Current or recent (within 30 days) exposure to any investigational drug.
* Patients having received a live vaccine within 28 days of study enrollment.
* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100,000/mm
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 2.5 x Upper Limit of Normal
* Patients with anaphylaxis and/or known allergic reactions to ACTH
* Previous Treatment with ACTH
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Concomitant or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of psychiatric disorder that would interfere with normal participation in this protocol.
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease).
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication.
* Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, PhD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Acthar (ACTH) Gel: Injected does of 80 units subcutaneously twice weekly for 6 months.
  Acthar (ACTH) Gel: Injected dose of 80 units subcutaneously twice weekly for 6 months.
Period: Overall Study
Arm/Group | Acthar (ACTH) Gel
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | ACTH Gel
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Complete or Partial Response to Treatment
Description: A complete response is defined by <300 mg proteinuria/24 hours and no greater than a 10% reduction in glomerular filtration rate (GFR) as determined by quantified creatinine clearance.
  A partial response is defined by >50% reduction in 24 hour proteinuria and no greater than a 25% reduction in baseline GFR as quantified creatinine clearance.
  No response is defined by < or equal to 50% reduction, unchanged or increasing proteinuria over baseline levels and a greater than a 25% reduction in baseline GFR as quantified creatinine clearance.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- Acthar (ACTH) Gel: Injected does of 80 units subcutaneously twice weekly for 6 months.
  ACTH (Acthar) Gel: Injected dose of 80 units subcutaneously twice weekly for 6 months.
Arm/Group | Acthar (ACTH) Gel
Number analyzed (Participants) | 19
Participants | 8

2. Secondary Outcome: Number of Subjects to Develop an Infection
Description: The number of subjects with infections was defined as the development of pneumonia or complicated urinary tract infection/Pyelonephritis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar (ACTH) Gel
Number analyzed (Participants) | 19
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from baseline until the completion of the final study visit for each subject, approximately 12 months.
Arm/Group | ACTH Gel
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 10/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTH Gel (N=19)
Infection (Infections and infestations) | 6 (6)
Acne (General disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Soreness (General disorders) | 1 (1)
Anxiety (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT02282930/Prot_SAP_000.pdf